CLINICAL TRIAL: NCT04506021
Title: A Multicenter Real World Study on Clinical Efficacy of Sodium Bicarbonate Ringer's Solution in Children With Biliary Atresia
Brief Title: A Real World Study on Clinical Efficacy of Bicarbonate Ringer's Solution in Biliary Atresia Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, J.X. Feng, prof., Tongji Hospital
Other Study IDs: TJH-MCTBR
Record Dates: First submitted 2020-08-03; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Biliary Atresia
Keywords: Biliary Atresia; Bicarbonate Ringer's solution; Perioperative fluid management
MeSH Terms: conditions — Biliary Atresia | interventions — glutathione-bicarbonate-Ringer solution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bicarbonate Ringer's Solution: According to the choices of the patients' immediate family members, patients will be divided into Bicarbonate Ringer's Solution.
  drug dosage form: Solution, Intravenous infusion. the drug dosage frequency and duration were no intervention
  Interventions: Drug: Bicarbonate Ringer's solution
- Other Crystalloid: According to the choices of patients' immediate family members, patients will be divided into Other Crystalloid.
  drug dosage form: Solution, Intravenous infusion. the drug dosage frequency and duration were no intervention
  Interventions: Drug: Other Crystalloid

INTERVENTIONS:
Drug: Bicarbonate Ringer's solution — According to the choices of the patients' immediate family members, patients will be divided into Bicarbonate Ringer's Solution. no Intervention.
  Groups: Bicarbonate Ringer's Solution
Drug: Other Crystalloid — According to the choices of the patients' immediate family members, patients will be divided into other clinical used crystalloid. no Intervention.
  Groups: Other Crystalloid

SUMMARY:
In most babies with biliary atresia (BA) bile ducts on the inside and outside of the liver are affected eventually leading to a complete blockage of bile flow from the liver. This in turn causes scarring (fibrosis) in the liver. The surgery called the Kasai procedure and eventually, a liver transplant could treat biliary atresia. However, children with BA have poor liver function, poor renal reserve, and poor ability to regulate water and electrolytes. Therefore, A reasonable and effective perioperative fluid management is more significant. Considering the high chlorine of saline, the liver burden of Lactated Ringer's solution and Acetated Ringer's solution, the Bicarbonate Ringer's solution which composition is similar to plasma, could be the best choice for perioperative fluid management of BA children. Therefore, we hypothesize that compared with other crystalloids, Bicarbonate Ringer's solution is a better choice to maintain water, electrolyte and acid-base balance in BA children.

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed with biliary atresia before surgery.
2. age less than 90 days.
3. American Society of Anesthesiologists score of 1~2.

Exclusion Criteria:

1. patients with severe allergies.
2. patients with severe deformities or lesions.
3. other situations not suitable for enrollment judged by researchers.

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study Population was diagnosed with biliary atresia, who need Intravenous infusion.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Arterial blood gas changes | 1 day
  Compared with the baseline, the patient's base excess and pH changes at the operation 1h, operation 2h, and the end of the operation.
Intraoperative dosage of sodium bicarbonate injection | 1 day
  Patients with acidosis during the operation needs to be corrected with sodium bicarbonate injection. We collect the amount of sodium bicarbonate injection used to correct metabolic acidosis during the operation
Chlorine concentration | 3 days
  We collected the concentration of chloride ion in the patient's blood and urine during the baseline, the operation and three days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Jiexiong Feng, Principal Investigator — Tongji hospital of huazhong university of science and technology